CLINICAL TRIAL: NCT01844921
Title: High Resolution Optical Imaging of the Esophagus Using the NvisionVLE™ Imaging System
Brief Title: High Resolution Optical Imaging of the Esophagus Using the Nvision Volumetric Laser Endomicroscopy (VLE™) Imaging System
Status: Completed | Type: Observational
Sponsor: NinePoint Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: 12_02
Record Dates: First submitted 2013-04-22; First posted 2013-05-03 (Estimated); Last update posted 2013-05-17 (Estimated); Status verified 2013-05

CONDITIONS: Undergoing Esophagogastroduodenoscopy (EGD)

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a single center, single arm, open label observational trial of patients undergoing EGD. The primary objective of this clinical trial is to evaluate the ability of physicians to position the NvisionVLE catheter to acquire an image of an area of the esophagus to identify and discriminate abnormal areas of tissue from normal.

ELIGIBILITY:
Inclusion Criteria:

* Males and females over the age of 18 years.
* Patients presenting for an EGD.
* Ability to provide written, informed consent.
* Females who are able to become pregnant, and are willing to take a pregnancy test.

Exclusion Criteria:

* Patients on anticoagulation undergoing high risk procedures in accordance to American Society For Gastrointestinal Endoscopy (ASGE) guideline for the management of antithrombotic agents for endoscopic procedures (2009)*.
* Patients with esophageal varices that preclude biopsies.
* Presence of an esophageal mass that precludes full distention of the balloon from the NvisionVLE Catheter.
* Patients with esophageal strictures that would prevent adequate expansion of the balloon from the NvisionVLE Catheter.
* Patients with known inflammatory disease, esophageal tears or ulcers, which would prohibit full distention of the balloon from the NvisionVLE Catheter.
* Patients with known eosinophilic esophagitis.
* Patients that are pregnant.
* Patients with a history of hemostasis disorders**.

  * Patients on anticoagulation undergoing low risk procedures are not excluded. **Hemostasis disorders will include, but will not be limited to: patients with hemophilia or other congenitally acquired clotting factor deficiencies, patients with cirrhosis with coagulopathy, patients known to have thrombocytopenia (<100,000 plt/ul) and individuals with von Willibrand's disease or other known platelet malfunction disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Males and females >18 years of age undergoing esophagogastroduodenoscopy (EGD).
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2013-04; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
The primary endpoint will be the number of patients achieving a VLE (volumetric laser endomicroscopy) image that includes stomach, gastro esophageal junction (GEJ) and esophagus. | Day of procedure
  Achieving a VLE image is defined as completing a full 6cm scan. This will be presented as a percentage of patients.

SECONDARY OUTCOMES:
The evaluation of procedural workflow and physician interface to the NvisionVLE Imaging Console. | Day of procedure.
  Procedural workflow and physician interface to the console will be assessed by a questionnaire that will be completed by the investigational staff involved in the procedure (eg - Were you (physician) able to position the catheter in the desired position?).

CONTACTS AND LOCATIONS:
Overall Officials: John Poneros, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States